CLINICAL TRIAL: NCT03704038
Title: Electrical Impedance Tomography Guided Assessment of Optimum PEEP Levels During Mechanical Ventilation in Lateral Decubitus Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Andrej Šribar, Specialist in anesthesiology and intensive are medicine, Principal Investigator, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018EIT
Record Dates: First submitted 2018-09-24; First posted 2018-10-12 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Mechanical Ventilation; Bioelectrical Impedance
Keywords: PEEP; Electrical impedance tomography; Mechanical ventialtion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PEEP 5 (Active Comparator)
  Interventions: Procedure: PEEP level
- PEEP 0 (Active Comparator)
  Interventions: Procedure: PEEP level
- PEEP 10 (Experimental)
  Interventions: Procedure: PEEP level

INTERVENTIONS:
Procedure: PEEP level — Patients will have variable PEEP levels and will be monitored

SUMMARY:
Goal of this study is to determine optimal PEEP levels for patients undergoing surgery in lateral decubitus position. Patients will be randomized into 3 groups - PEEP 0, 5 and 10 mbar. Endotracheal anesthesia will be conducted with propofol, fentanyl, rocuronium and sevoflurane/O2/air gas mixture.

Patients with preexisting lung disease, organ transplants and disseminated malignant disease will be excluded.

Demographic data - age, weight, height, ASA status, smoking history will be recorded. EIT measured parameters - tidal variation ratio of nondependent and dependent lung, regional end-tidal and end-expiratory lung impedances as well as horizontal and vertical centers of ventilation will be recorded and calculated at 3 time points - before anesthesia induction, 5 minutes after lateral positioning of the patient and 90 minutes after lateral positioning. ABGs will be sampled to calculate aA gradient and Horovitz quotient at those time points as well as measured hemodynamic parameters (HR, BP, CI, SVI).

Primary endpoints for the study are nondependent/dependent tidal variation ratios measured at predefined time points and changes in ABGs. Secondary endpoints are number of postoperative pulmonary complications (defined as new onset of pneumonia during 28 days of followup), length of hospital stay and changes in hemodynamic parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for nephrectomy, adrenalectomy or urterotomy surgery which will be performed in lateral decubitus position
* signed informed consent form

Exclusion Criteria:

* preexisting moderate to severe obstructive (GOLD score > 1) or restrictive lung disease (FVC < 85%)
* history of organ transplant
* disseminated malignant disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change of nondependent / dependent tidal variation | Baseline, 10 and 90 minutes post lateral positioning
  Measured by EIT

SECONDARY OUTCOMES:
Change of a-A gradient | Baseline, 10 and 90 minutes post lateral positioning
  Measured by ABG analysis
Duration of hospital stay | Up to 28 days
  Between groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Šribar, MD, PhD, Principal Investigator — Anesthesiologist and Critical Care specialist
Locations (1):
- University Hospital Dubrava, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No